CLINICAL TRIAL: NCT06256900
Title: Flow Controlled Ventilation to Improve Postoperative Pulmonary Outcome After Robot-assisted Laparoscopic Surgery - a Prospective, Randomised, Single-blinded, Controlled and Single-centre Investigation
Brief Title: Flow Controlled Ventilation in Robot-assisted Laparoscopic Surgery
Acronym: FCV-IMPALA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The preparation and execution of this study were discontinued due to a range of practical constraints. Including logistical and operational challenges that would have compromised the study's feasibility and effective and questioning reliable results.
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Dr. Timur Yurttas, Principal Investigator, Senior Physician Anesthesiology, MD, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-02285
Record Dates: First submitted 2024-01-29; First posted 2024-02-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-08

CONDITIONS: Mechanical Ventilation Complication; Postoperative Pulmonary Atelectasis
Keywords: Flow-controlled ventilation; Postoperative pulmonary complications; electrical impedance tomography
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-center study
Who Masked: Participant
Masking Description: single blinded to the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flow-controlled ventilation (Experimental): Experimental intervention FCV (EVONE, Ventinova Medical): PEEP and Peak inspiratory pressure titration guided by dynamic compliance.
  Interventions: Other: Flow-controlled ventilation
- Pressure-controlled ventilation (Active Comparator): Control intervention PCV (Dräger Medical, Atlan A350): lung-protective ventilation to current best practice. Settings determined by the attending anesthesiologist (based on the internal SOP: intraoperative ventilation in robot-assisted laparoscopic surgery).
  Interventions: Other: Pressure-controlled ventilation

INTERVENTIONS:
Other: Flow-controlled ventilation — FCV mode during robot-assisted laparoscopic surgery
  Other Names: FCV
  Arms: Flow-controlled ventilation
Other: Pressure-controlled ventilation — PCVmode during robot-assisted laparoscopic surgery
  Other Names: PCV
  Arms: Pressure-controlled ventilation

SUMMARY:
The optimization of ventilation is especially important during general anaesthesia, when active, physiologic respiration suspends and is replaced by non-physiologic mechanical positive pressure ventilation. Aiming at preserving compliance of lung tissue to guarantee an effective gas exchange is to avoid an excessive pressure application, especially in extreme positioning of the patient (Trendelenburg positioning) and/or pneumoperitoneum resulting in additional non-physiologic intrathoracic pressure. Perioperative lung protection strategies have steadily improved in recent years to reduce complications from mechanical ventilation, but postoperative pulmonary complications remain a risk factor for increased morbidity and mortality.

DETAILED DESCRIPTION:
Mechanical ventilation is crucial during general anesthesia, with ongoing efforts to refine strategies for optimal respiratory support. Important articles on perioperative ventilation explored key aspects, including PEEP application, tidal volume effects, PPC after major surgeries, and perioperative oxygen titration to mitigate oxidative stress. PEEP plays a pivotal role in enhancing oxygenation and preventing atelectasis during mechanical ventilation. Landmark studies by the ARDS Network highlight the importance of customizing PEEP application. This tailored approach not only improves respiratory mechanics but also reduces the risk of barotrauma, underscoring the crucial impact of personalized PEEP strategies. Concurrently, adopting a lung-protective strategy with low tidal volumes, has proven effective in mitigating ventilator-induced lung injury. These strategies aim to strike a balance between optimal oxygenation and minimizing potential complications associated with mechanical ventilation. Despite advancements in perioperative care, PPC remain a concern, particularly following major surgical procedures. Recent investigations emphasize the multifactorial nature of these complications. Early identification of risk factors and meticulous monitoring are crucial to reducing the incidence of complications such as atelectasis, pneumonia, and respiratory insufficiency. Understanding the interplay between mechanical ventilation strategies and postoperative outcomes is essential for improving patient recovery. The pursuit of optimal oxygenation must be balanced against the potential for oxygen toxicity and oxidative stress. Available studies shed light on the delicate equilibrium required in maintaining adequate oxygen delivery while avoiding the detrimental effects of hyperoxia. Clinicians must consider individual patient factors and tailor oxygen therapy to prevent oxidative stress, which can contribute to tissue damage and compromise overall patient well-being. FCV is a new ventilation strategy designed to minimize the mechanical effects of perioperative ventilation on lung tissue. Compared to traditionally employed ventilation strategies, gas flow is controlled during both inspiration and expiration in FCV. In particular, the almost linear pressure drop during the expiratory phase of FCV has been shown in various ex vivo/experimental and clinical studies to improve gas exchange and the proportion of ventilated lung tissue.

Ongoing advancements in mechanical ventilation shape anesthesia practices with a focus on evidence-based approaches for patient safety. Building on prior findings, this study explores the benefits of the novel ventilation approach, FCV, aiming to reduce dissipative energy and alveolar stress. The investigators hypothesize positive impacts on perioperative ventilation, vital parameters, and a decreased incidence of PPC, contributing to overall postoperative morbidity and mortality reduction.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective robot-assisted laparoscopic surgery (either abdominal, urologic or gynecologic surgery) with a duration of expected ventilation of ≥ 90 minutes
* Male or female aged ≥ 18 years
* ASA Physical Status Classification System score I - III
* Must be willing and able to give written informed consent to participate in the study and agree to comply with the study protocol prior to initiation of any study-mandated procedure and study intervention

Exclusion Criteria:

* Patient with weight < 40 kg ideal body weight
* ASA Physical Status Classification System score IV - VI
* Previous enrolment into the current study
* Enrolment of study investigator, his/her family members, employees and other dependent persons
* If female and of childbearing potential: known pregnancy or a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Differences in the number of patients developing postoperative pulmonary complications | to postoperative day 5/discharge
  Development of PPC (composite endpoint including pneumonia, bronchospasm, atelectasis, pulmonary congestion, respiratory failure, pleural effusion, pneumothorax, requirement for mechanical ventilation) within the first 5 postoperative days (or until discharge).
  * Constant postoperative monitoring of clinical features indicating PPC
  * EIT parameters indicating atelectasis (defined by EIT derived parameters Global Inhomogenity Index, Tidal Impedance Variation, end-expiratory lung impedance) measurement after arrival at the PACU.
  * Requirement of additional oxygen will be evaluated after transfer to the PACU/ICU. Air test indicating additional oxygen requirement, SpO2 <90% / <88% in case of risk of hypercapnic respiratory failure.
  * If unplanned and continued mechanical ventilation is required after surgery this will count as fulfilled primary endpoint.

SECONDARY OUTCOMES:
Differences in Clara-Cell 16 serum concentrations | periprocedural
  Presence and increase of blood biomarkers indicating alveolar shear stress compared between groups. Blood samples will be required to determine CC16 (3x during the course of the study, approx. 5ml blood each).
  * Baseline (during preoperative anaesthesia consultation or during preparations before induction of anaesthesia
  * During intervention: ca. 60 minutes after final adjustments of Trendelenburg positioning/pneumoperitoneum
  * After transfer to PACU/ICU respectively
Differences in area under the curve of postoperative modified Horovitz index | first hour after surgery
  maximal area under the curve of SpO2/FiO2 compared between groups during first hour after surgery/arrival at the PACU. Derived from data recorded in the electronic anesthesia protocol.
Differences in end-tidal to capillary/arterial CO2 gradient | periprocedural
  Maximal end-tidal to capillary/arterial CO2 gradient compared between groups. (Capillary blood gases can accurately reflect arterial pH, pCO2 and Hb. Because arterial cannulation is not mandatory in the patient population, the investigators choose to determine the end-tidal to arterial CO2 gradient by assessing capillary blood gas, which has been shown to accurately reflect arterial CO2). Derived from data recorded in the electronic anesthesia protocol.
Differences in minimal required intraoperative FiO2 concentration | periprocedural
  Minimal required intraoperative FiO2 to ensure an adequate perioperative oxygenation (defined as min. oximetric SpO2 of >94%). Derived from data recorded in the electronic anesthesia protocol.
Differences in parameters derived from the electrical impedance tomography | periprocedural
  Comparison of spatial and regional ventilation patterns during intervention between groups. Comparison of respiratory system compliacen, end-expiratory lung volume between groups at baseline (before surgical procedures in supine position), during intervention (ca. 60 min after Trendelenburg/pneumoperitoneum) and after return to supine position/end of pneumoperitoneum.
  Whether FCV has an influence on parameters visualized and measured by EIT, these data will be monitored and evaluated during (secondary outcome assessment) and after (primary outcome assessment) the intervention (measurements at: baseline - during intervention (60min after Trendelenburg/Pneumoperitoneum) - after Trendelenburg/Pneumoperitoneum - after arrival at PACU)
Differences in perioperative ventilation/oxygenation parameters | periprocedural
  Differences in perioperative ventilation and oxygenation parameters (minimal FiO2, min/max. PEEP, min/max. compliance), compared between groups. Data derived from the electronic anesthesia protocol.

OTHER OUTCOMES:
Number of patients developing events defined as safety events | periprocedural
  Determine number of patients with potential ventilation-related complications in the perioperative setting, which are not causally related to the surgical procedure and require a change in ventilation technique ((i.e., conversion from FCV to PCV/VCV; or conversion from PCV to VCV) in order to guarantee patient safety (based on sufficient oxygenation or sufficient elimination of CO2, respectively, and the decision of the responsible anesthesiologist). Further, the safety objective is to assess the occurrence of intervention-related serious adverse events.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code